CLINICAL TRIAL: NCT01511601
Title: Apheresis to Obtain Plasma and Leukocytes in Mali for In Vitro Studies
Brief Title: Apheresis to Obtain Plasma and White Blood Cells in Malies
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912048; 12-I-N048
Record Dates: First submitted 2012-01-13; First posted 2012-01-18 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-07-28

CONDITIONS: Malaria
Keywords: Apheresis; Leukocytes; Plasma; Plamodium Falciparum Malaria; Immunology
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Some clinical trials require larger amounts of plasma and white blood cells than can be collected through simple blood donations. Apheresis is a procedure used to collect parts of the blood for study and return the rest of the blood to the donor. Healthy volunteers who provide plasma and white blood cells for study may need to give multiple donations. Researchers want to use apheresis to collect plasma and white blood cells from healthy volunteers in Mali.

Objectives:

- To collect plasma and white blood cells from healthy volunteers in Mali.

Eligibility:

* Healthy volunteers between 18 and 55 years of age.
* Volunteers must be in National Institute of Allergy and Infectious Diseases clinical trials.

Design:

* Participants will be screened with a physical exam and medical history. They will also provide basic blood and urine samples.
* Participants will have apheresis to collect plasma and white blood cells for study. Before each collection, they will provide a small blood sample for testing. They will be monitored during and after donation to prevent side effects.
* Under this protocol, participants may have apheresis up to six times per year.
* No treatment will be provided as part of this protocol....

DETAILED DESCRIPTION:
To carry out in vitro research procedures on plasma or leukocyte components of whole blood, it is often necessary to obtain larger quantities of plasma or leukocytes than can be safely obtained by simple phlebotomy. These components can be easily and safely obtained using a well-established standard apheresis procedure that is in common use at the National Institutes of Health Apheresis Unit. This protocol describes the implementation of the same apheresis procedure at the National Blood Transfusion Center in Bamako, Mali. This is not a research protocol per se, but rather an adjunct protocol which allows healthy donors 18-55 years of age to undergo apheresis. Subjects must already be enrolled in another protocol which has been approved by the National Institute of Allergy and Infectious Diseases Institutional Review Board and the Faculty of Medicine, Pharmacy, and Odonto-Stomatology Ethics Committee.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals 18-55 years of age are eligible to enter the study if they:

* Are enrolled on another NIAID/FMPOS-approved protocol.
* Weigh greater than or equal to 50 kg.
* Agree to have blood specimens stored for future studies.
* Agree to undergo genetic testing.
* Agree to undergo HIV, hepatitis B, and hepatitis C virus testing.

EXCLUSION CRITERIA:

The following criteria are exclusionary:

* Positive at screening for HIV, hepatitis B, and/or hepatitis C.
* Cardiovascular instability (blood pressure <90/50 or >180/100; pulse <40 or >110.
* Inadequate peripheral venous access.
* Anemia (hemoglobin <11 g/dL).
* Current use of corticosteroids or other immunosuppressants.
* Underlying heart disease, lung disease, bleeding disorder, or other conditions that, in the judgment of the investigator, contraindicates apheresis.
* Temperature greater than or equal to 37.5 degree C or other clinical evidence of an acute infection.
* Currently pregnant or breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12-20; Study Completion 2016-07-28

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Crompton, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)